CLINICAL TRIAL: NCT04852523
Title: Assessing the Value of 18F-Fluciclovine PET/CT in the Assessment of Pancreatic Transplants
Brief Title: 18F-Fluciclovine PET/CT in the Assessment of Pancreatic Transplants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeffrey Yap, PhD, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 136948
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pancreatitis, Graft; Pancreatic Transplant Post-Transplant Dysfunction Rejection
MeSH Terms: conditions — Pancreatitis, Graft | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 18F fluciclovine Administration (Experimental): * Initial normal standardized uptake values (SUV) of the pancreas, liver, and blood pool will be obtained from 50archived previous 18F-Fluciclovine studies, as there are no normal ranges in the literature. This will be done by retrospective medical record review after a waiver of consent/authorization is obtained from the local IRB.
  * Informed consent will be obtained from 10 patients with pancreatic allografts, and each will undergo an 18F-Fluciclovine study. These patients will not be suspected of having current rejection or allograft dysfunction. Timing of 18F-Fluciclovine PET/CT scans will be planned to coincide with standard-of-care imaging studies and laboratory tests.
  * The 18F-Fluciclovine study will be compared with the patients' standard-standard-of-care US and/or CT with the assessment of ease of visualization of the pancreatic allograft.
  Interventions: Drug: 18F-fluciclovine

INTERVENTIONS:
Drug: 18F-fluciclovine — 18F-Fluciclovine is a synthetic L-leucine amino acid used clinically for PET imaging in patients with biochemical recurrence of prostate cancer following definitive therapy. The pancreas accumulates striking amounts of Axumin, where it is considered a normal finding. Pancreatic beta-cell function may be slow to recover following pancreatic transplantation and may vary as a function of perioperative steroid administration, acute rejection, inadequate islet cell transplantation, allograft pancreatitis or compromised blood supply. Viability of the allograft is a common clinical concern and is difficult to assess based on insulin, C-peptide, and blood sugar levels. Rapid identification of compromised allograft viability is critical in the management of these patients.
  Other Names: Axumin

SUMMARY:
Hypothesis 1: 18F-Fluciclovine PET/CT can correctly and easily identify the pancreatic allograft and determine its viability

Aim 1: Assess whether 18F-Fluciclovine can identify the pancreatic allograft accurately and assess its viability and visibility

Hypothesis 2: 18F-Fluciclovine PET/CT uptake in the pancreas (SUV) is related to total pancreatic function and therefore can indicate whether the pancreatic allograft is at risk of rejection

Aim 2: Assess whether 18F-Fluciclovine uptake in the pancreas can be a surrogate for pancreatic function

DETAILED DESCRIPTION:
18F-Fluciclovine is a synthetic L-leucine amino acid used clinically for PET imaging in patients with biochemical recurrence of prostate cancer following definitive therapy. The pancreas accumulates striking amounts of Axumin, where it is considered a normal finding. Pancreatic beta-cell function may be slow to recover following pancreatic transplantation and may vary as a function of perioperative steroid administration, acute rejection, inadequate islet cell transplantation, allograft pancreatitis or compromised blood supply. The viability of the allograft is a common clinical concern and is difficult to assess based on insulin, C-peptide, and blood sugar levels. Rapid identification of compromised allograft viability is critical in the management of these patients.

Pancreas transplants are usually assessed via ultrasound as a first-line modality. However, visualization is largely obscured due to the intraperitoneal location of the transplant. There is often overlying gas and due to the depth of the transplant, there is poor visualization with ultrasound. Additionally, the transplant lacks a capsule

which results in its being ill-defined and difficult to distinguish from adjacent structures. Computed tomography can also be used to assess pancreas transplants, however, most transplant patients often have concurrent renal transplants which limits the use of intravenous iodinated contrast. On non-contrast CT, it can be difficult to assess and distinguish the pancreas transplant from the adjacent bowel. Magnetic Resonance Imaging (MRI) can be useful and has better soft-tissue contrast compared to CT. However, it has a similar issue with regards to limited intravenous gadolinium contrast administration due to concurrent renal transplant in this group of patients. In all three modalities, there is no functional assessment of the allograft and whether there is still appropriate pancreatic function.

This is the reason for our proposed study, given that 18F-Fluciclovine is readily taken up by the pancreas and it would help radiologists readily identify where the allograft is located, whether it is viable, and whether there is a normal function of the allograft. It should be noted that leucine serves both as a fuel, as well as in a regulatory capacity for pancreatic beta-cell function. However, uptake of 18F-Fluciclovine in the pancreas is not likely to be specific for beta-cell function since acinar cell function requires L-amino acids. However, overall pancreatic viability is relevant to both acinar cell and beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

* 18 or over in age
* Have any type of pancreatic transplant
* Able to consent for 18F-Fluciclovine PET/CT scan
* For archived 18F-Fluciclovine PET/CT scan reviews, only scans of non-diabetic patients will be included.

Exclusion Criteria:

- Patient with known prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Measurement of Pancreatic Allograft Viability after 18F-Fluciclovine Utilization | This outcome will be measured after the radiologic images have been processed and archived (within 24 hours of intervention) and laboratory results are certified (within 24 hours of intervention).
  Regions of Interest (ROI) will be placed on the pancreas to determine the standardized uptake value (SUV) which requires the correlation of the patient's standard of care laboratory results. A higher SUV result would indicate stronger viability for the allograft.
Measurement of Pancreatic Allograft Visibility after 18F-Fluciclovine Utilization | These reviews will take place within 72 hours of the radiologic imaging taking place for each participant.
  Pancreatic allograft visibility after the use of 18F-Fluciclovine will be measured by 3 separate nuclear medicine/ radiology readers. Each reviewer will grade the images on a scale from 1 to 5, 5 being the most visible when compared to the non-contrast CT images.
Measurement of Pancreatic Allograft Uptake after 18F-Fluciclovine Utilization | This outcome will be measured after the radiologic images have been processed and archived (within 72 hours of intervention).
  Regions of Interest (ROI) will be placed on the pancreas to determine the standardized uptake value (SUV). A higher SUV result will indicate a higher likelihood that allograft rejection is not/will not take place.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided